CLINICAL TRIAL: NCT05293288
Title: EEG-guided General Anesthesia vs. Routine Care and Cumulative Dose of Norepinephrine in Patients Having Vascular Surgery: a Pilot Randomized Trial
Brief Title: Effect of EEG-guided General Anesthesia on Cumulative Dose of Norepinephrine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Kristen Thomsen, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-10155-BO-ff
Record Dates: First submitted 2022-03-03; First posted 2022-03-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EEG-guided general anesthesia (Experimental): EEG-guided general anesthesia group (i.e., intervention group): For pEEG monitoring we will use the SEDLine monitor (Masimo, Irvine, CA) which provides the patient state index (PSi; a processed EEG parameter with values from 1 to 100), density spectral array (DSA; a display that represents the frequencies and amplitudes of brain waves through time), spectral edge frequency (SEF), and the raw EEG signal.
  Interventions: Device: EEG-guided general anesthesia
- Routine care (No Intervention): Routine care group (i.e., control group): Adjustment of depth of general anesthesia will be at the discretion of the treating anesthesiologist.

INTERVENTIONS:
Device: EEG-guided general anesthesia — pEEG monitoring will start with the beginning of induction of general anesthesia and will end with the end of surgery (surgical suture). In the EEG-guided group, depth of anesthesia will be adjusted to target PSI values between 25 and 50 and spectral edge frequency between 10 and 15. In case of contradictory values, the raw EEG waveforms, ARTF, EMG, as well as the overall clinical situation will be evaluated for decision making.
  Arms: EEG-guided general anesthesia

SUMMARY:
Intraoperative hypotension is common in patients having non-cardiac surgery under general anesthesia and is associated with major postoperative complications including myocardial injury, AKI, and death.

Intraoperative hypotension is also common in patients having vascular surgery. To treat intraoperative hypotension, vasopressors - such as norepinephrine - and fluids are used. However, high-dose vasopressor and excessive fluid therapy are also associated with postoperative complications.

The depth of general anesthesia may be a modifiable cause of intraoperative hypotension. Deep levels of general anesthesia may cause cardiovascular depression with intraoperative hypotension and higher vasopressor requirements. Optimal depth of general anesthesia is defined as a state in which the patient is at low risk of recall of intraoperative events while maintaining blood pressure stability with minimal intervention.

Depth of anesthesia can be confirmed using clinical signs, the concentration of inhaled or intravenous anesthetics, or neuromonitoring such as processed electroencephalography (pEEG). pEEG presents an opportunity to monitor changes in human brain electrical activity and to help estimating the patients' level of (un)consciousness and the optimal depth of anesthesia. EEG-guided general anesthesia may thus decrease norepinephrine doses needed to treat intraoperative hypotension in patients having surgery.

ELIGIBILITY:
We will include consenting patients ≥45 years scheduled for elective vascular surgery under general anesthesia if:

* surgery is expected to last at least 60 min AND
* the estimated blood loss during surgery is less than 1000 mL AND
* intraarterial blood pressure monitoring (arterial catheter) is planned during surgery

We will not include patients with previous transplantation of kidney, liver, heart, or lung and those who are septic (according to current Sepsis-3 definition). And we will not include patients with American Society of Anesthesiologists' physical status V and VI, or pregnancy.

We will exclude patients after randomization if they were treated with vasopressors others than norepinephrine during surgery.

Written informed consent will be obtained from all patients prior to study inclusion.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Cumulative norepinephrine dose | Outcome meassure will be assessed at the end of surgery
  Time-weighted cumulative norepinephrine dose normalized to the patient's actual body weight: cumulative norepinephrine dose [µg] / body weight [kg] / length of surgery [min]; unit: µg/kg/min

SECONDARY OUTCOMES:
Incidence and severity of intraoperative hypotension | Outcome meassure will be assessed at the end of surgery
  Cumulative minutes below MAP of 65 mmHg
Incidence and severity of intraoperative hypotension | Outcome meassure will be assessed at the end of surgery
  Area under a mean arterial pressure of 65 mmHg
Incidence and severity of intraoperative hypotension | Outcome meassure will be assessed at the end of surgery
  Time-weighted average MAP under 65 mmHg
Hospital length of stay | Through study completion, an average of 1 year
  Hospital length of stay
ICU length of stay | Through study completion, an average of 1 year
  ICU length of stay
Hospital mortality | Through study completion, an average of 1 year
  Hospital mortality

OTHER OUTCOMES:
Postoperative AKI | 30 days before the surgery until the first 7 postoperative days
  Postoperative AKI defined as an increase in serum creatinine concentration of ≥0.3 mg/dL within any 48 h period within 7 postoperative days or of ≥50% from baseline within the first 7 postoperative days (based on: Kidney Disease: Improving Global Outcomes (KDIGO) Clinical Practice Guideline for Acute Kidney Injury. The preoperative baseline serum creatinine concentration will be defined as the most recent recorded measurement within 30 days before the surgery. We will consider AKI as a binary outcome (no AKI vs. AKI of any stage). We will consider serum creatinine values when measured per routine care.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomsen KK, Sessler DI, Krause L, Hoppe P, Opitz B, Kessler T, Chindris V, Bergholz A, Flick M, Kouz K, Zollner C, Schulte-Uentrop L, Saugel B. Processed electroencephalography-guided general anesthesia and norepinephrine requirements: A randomized trial in patients having vascular surgery. J Clin Anesth. 2024 Aug;95:111459. doi: 10.1016/j.jclinane.2024.111459. Epub 2024 Apr 9. PMID 38599161